CLINICAL TRIAL: NCT02533726
Title: Randomized Control Trial Evaluating Optimal Patient Turning Procedures for Reducing Hospital Acquired Pressure Ulcers
Brief Title: Optimal Patient Turning for Reducing Hospital Acquired Pressure Ulcers
Acronym: LS-HAPU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Leaf Healthcare, Inc. (Industry)
Responsible Party: Principal Investigator, David Pickham, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 33144
Record Dates: First submitted 2015-08-17; First posted 2015-08-27 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2017-09

CONDITIONS: Pressure Ulcer
Keywords: Bed Sores; Bedsores; Decubitus Ulcer; Pressure Sore
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment - Optimal Turning (Experimental): All patients will have a sensor applied. Patients within this arm will receive care from nurses who have access to a User Dashboard that provides visual advisories for patient turning, based on data obtained from a wearable patient sensor (Leaf Healthcare, Inc.).
  Interventions: Other: Optimal Turning; Other: Patient Sensor
- Control - Standard Care (Active Comparator): All patients will have a sensor applied. Patients within this arm will receive care from nurses who DO NOT have access to a User Dashboard that provides visual advisories for patient turning. Instead, these patients will receive standard care practices, patient turning initiated by nurses as necessary.
  Interventions: Other: Standard Care Practices; Other: Patient Sensor

INTERVENTIONS:
Other: Optimal Turning — Patients within this arm will receive optimal turning practices. Nurses caring for these patients will receive real-time quantitative measures of patient turning procedures from the User Dashboard and provide a visual advisory to the nurse for the time to next turn.
  Other Names: Patient Turning; Pressure Ulcer Prevention
  Arms: Treatment - Optimal Turning
Other: Standard Care Practices — Patients within this arm will receive standard preventative care practices - that is, nurses will provide standard care as necessary, without the aid of visual advisories from a patient sensor.
  Arms: Control - Standard Care
Other: Patient Sensor — A small sensor with adhesive backing is applied to the upper chest (midline) of the patient. Sensor tracks and records body movement and position, and displays this on a User Dashboard located on a computer at the bedside.
  Other Names: Leaf Healthcare Patient Monitoring Sensor

SUMMARY:
The purpose of this study is to test whether optimal patient turning, strictly every 2 hours with at least 15 minutes of tissue decompression, reduces the occurrence of hospital acquired pressure ulcers.

DETAILED DESCRIPTION:
This single site, open label, two arm randomized control trial aims to evaluate whether optimal patient turning, strictly every 2 hours with at least 15 minutes of tissue decompression, reduces the occurrence of hospital acquired pressure ulcers. Optimal turning procedures will be obtained with the use of a patient monitoring system (Leaf Healthcare, Inc.) and compared to standard preventative care practices.

Sensors were placed on all participants as they were admitted to ICU. A nurse's user dashboard was turned on for participants in the Optimal Turning Group, but was not turned on for participants in the Standard Care group.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age)
* Admission to Intensive Care Unit

Exclusion Criteria:

* Children (<18 years of age)
* Adhesive allergy
* Physical limitation for sensor application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pickham, PhD, Principal Investigator — Stanford Health Care
Locations (1):
- Stanford Health Care, Stanford, California, United States

REFERENCES:
- [Derived] Pickham D, Ballew B, Ebong K, Shinn J, Lough ME, Mayer B. Evaluating optimal patient-turning procedures for reducing hospital-acquired pressure ulcers (LS-HAPU): study protocol for a randomized controlled trial. Trials. 2016 Apr 6;17:190. doi: 10.1186/s13063-016-1313-5. PMID 27053145

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment - Optimal Turning: All patients had a sensor applied. Patients within this arm received care from nurses who had access to a User Dashboard that provided visual advisories for patient turning, based on data obtained from the wearable patient sensor.
- Control - Standard Care: All patients had a sensor applied. Patients within this arm received care from nurses who did not have access to a User Dashboard that provided visual advisories for patient turning. Instead, these patients received standard care practices, patient turning initiated by nurses as necessary.
Period: Initial Allocation
Arm/Group | Treatment - Optimal Turning | Control - Standard Care
Started | 659 | 653
Completed | 659 | 653
Not Completed | 0 | 0
Period: Treatment
Arm/Group | Treatment - Optimal Turning | Control - Standard Care
Started (54 participants allocated to Standard Care actually received Optimal Turning) | 709 (54 participants allocated to Standard Care actually received Optimal Turning) | 603 (4 participants allocated to Optimal Turning actually received Standard Care)
Per Protocol Population (Met minimum monitoring period (>2h) and did not receive both interventions) | 671 | 555
Completed | 709 | 603
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Per protocol population according to treatment received (met minimum monitoring period (>2h) and did not receive both interventions)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment - Optimal Turning | Control - Standard Care | Total
Number analyzed (Participants) | 671 | 555 | 1226
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17) | 60 (18) | 60 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 253 | 551
  Male | 373 | 302 | 675
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 113 | 82 | 195
  Not Hispanic or Latino | 538 | 458 | 996
  Unknown or Not Reported | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Pressure Ulcer According to the National Pressure Ulcer Advisory Panel (NPUAP) Criteria for Pressure Ulcers
Description: NPUAP criteria include 4 stages and 2 unstaged criteria. The count of patients with pressure ulcer according to any of the criteria are reported.
  * Stage 1: Non-blanchable erythema of intact skin
  * Stage 2: Partial-thickness skin loss with exposed dermis
  * Stage 3: Full-thickness skin loss
  * Stage 4: Full-thickness skin and tissue loss
  * Unstageable: Obscured full-thickness skin and tissue loss
  * Suspected deep tissue injury: Persistent non-blanchable deep red, maroon or purple discoloration
Time Frame: Duration of ICU admission (average 1 week)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment - Optimal Turning | Control - Standard Care
Number analyzed (Participants) | 671 | 555
Participants | 5 | 15
Statistical Analysis 1: Comparison: Treatment - Optimal Turning vs Control - Standard Care; Per-protocol (PP) analysis, consistent with regulatory guidance (FDA); Test type: Superiority; p = .012, Fisher Exact; Odds Ratio (OR) = .27, 95% CI 2-sided [.1 to .75]
Statistical Analysis 2: Comparison: Treatment - Optimal Turning vs Control - Standard Care; Per protocol analysis adjusted for admitting team, unit of admission, and risk for pressure injury; Test type: Other; p = 0.015, Fisher Exact; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.06 to 0.74]

2. Secondary Outcome: Compliance With Patient Turning Procedures
Description: Compliance is reported as the percentage of time during ICU admission that patients received turning every two hours.
Time Frame: Duration of ICU admission (average 1 week)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Treatment - Optimal Turning | Control - Standard Care
Number analyzed (Participants) | 671 | 555
percentage of time | 67 (19.5) | 54 (22.3)

ADVERSE EVENTS:
Time Frame: Duration of ICU admission (average 1 week)
Description: Adverse events are reported according to treatment received
Arm/Group | Treatment - Optimal Turning | Control - Standard Care
Serious Adverse Events (participants affected / at risk) | 0/709 | 0/603
Other Adverse Events (participants affected / at risk) | 0/709 | 0/603

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No